CLINICAL TRIAL: NCT02317120
Title: BRCA1 and BRCA2 Mutation in Romanian Population: a Study of Genotype - Phenotype Correlation at Diagnosis With Prospective Disease Outcome and Survival
Status: Completed | Type: Observational
Sponsor: Alexandru Eniu (Other)
Collaborators: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor-Investigator, Alexandru Eniu, MD PhD, Prof. Dr. I. Chiricuta Institute of Oncology
Organization: Prof. Dr. I. Chiricuta Institute of Oncology (Other)
Other Study IDs: D0810C00088
Record Dates: First submitted 2014-12-11; First posted 2014-12-15 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: To Determine the Prevalence, Penetrance of BRCA1 and BRCA2 Mutations in Romanian Womens With Breast or Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Multiplex Polymerase Chain Reaction; monophosphoryl lipid A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Genetic: NGS BRCA 1 and BRCA 2 full sequencing
Genetic: Multiplex ligation-dependent probe amplification (MPLA) BRCA1 BRCA2 — Firstly many pairs of probes, containing: a universal primer sequence, a specific hybridisation target sequence and a stuffer DNA region to vary the size of the resulting product, are hybridised adjacent to each other on the target DNA strand .The two adjacent probe sequences are ligated to form a continuous section of DNA.The ligated probes are then amplified using PCR. The amplified fragments are analysed by capillary electrophoresis to detect the different fragment lengths. These data can be analysed to show the relative copy number of each fragment that is present in the sample.

SUMMARY:
Primary objective To determine BRCA1 and BRCA2 variants in 250 Romanian women with breast/ovarian cancer selected for likeliness to harbor germline mutations in these genes by specific criteria for high-risk status including age at disease onset.

Secondary objective Considering the fact that BRCA testing is not a routine procedure in Romania and mutation prevalence varies in different populations, we intend to look for the founder mutation in our population, running full BRCA genes sequencing to a representative population sample. This would allow a more targeted approach to real-life practice and would ensure personalized solutions for every patient in need.

ELIGIBILITY:
Inclusion Criteria:

Categories of patients to be recruited for complete sequencing of all BRCA1 and BRCA2 exons are subjects who have been diagnosed with breast or ovarion cancer and who are:

1)40 years of age or younger 2)Triple negative breast cancer diagnosed before 50 years of age 3)Male with breast cancer 4)Bilateral breast cancer, first tumor diagnosed before 50 years of age 5)2) + 50 years of age or younger with at least one (first degree) relative diagnosed with breast cancer at 50 years of age or younger or a first degree relative with ovarian cancer 6)of any age with 2 or more relatives with breast cancer 7)of any age with 2 or more relatives with ovarian cancer 8)of any age with a personal history of ovarian cancer, tuba or peritoneal carcinoma 9)Two patients in same branch of the family, Prostate ca < 60 yr and 1st degree relative with BC < 50 yr 10)Two or more 1st and 2nd degree relatives of a patient with breast cancer, at least one of them <50 yr 11)of any age with a family history of male breast cancer or are at increased risk of having a BRCA mutation based on BRCAPRO or Tyrer-Cuzick models

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Womens who have been diagnosed with breast/ovarian cancer , carriers of a high risk of gBRCA mutations based on prespecified inclusion criterias
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
BRCA1 and BRCA2 variants prevalence and penetrance at Romanian women with breast/ovarian cancer selected for likeliness to harbor germline mutations | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Eniu, MD,PhD, Study Director — ESMO
Locations (1):
- ChiricutaIO, Cluj-Napoca, Cluj Napoca, Romania